CLINICAL TRIAL: NCT00830401
Title: Comparative Controlled Trial of Treatment of Minor Unexpected Uterine Cavity Abnormalities Diagnosed by Office Hysteroscopy Screening in Women Indicated for IVF
Brief Title: The Impact of Treating Minor Uterine Cavity Abnormalities Diagnosed by Office Hysteroscopy in Unselected In Vitro Fertilization (IVF) Cases
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Abnormality prevalence revealed to be much lower than expected.
Sponsor: UMC Utrecht (Other)
Collaborators: AZ-VUB (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, Professor, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TEAtrial
Record Dates: First submitted 2009-01-26; First posted 2009-01-27 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Minor Intra-uterine Abnormalities
Keywords: intra-uterine abnormalities; intracavitary pathology; hysteroscopy; IVF; ICSI; polyp; myoma; adhesion; septum; endometritis
MeSH Terms: conditions — Polyps; Myoma; Tissue Adhesions; Endometritis | interventions — Ofloxacin; Doxycycline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): One or more of the predefined minor intra-uterine abnormalities have been detected, but not treated during hysteroscopy.
- 2 (Active Comparator): One or more of the predefined minor intra-uterine abnormalities have been detected and treated during hysteroscopy.
  Interventions: Procedure: Treatment of predefined abnormality by hysteroscopic surgery; Drug: Ofloxacinum/Doxycycline

INTERVENTIONS:
Procedure: Treatment of predefined abnormality by hysteroscopic surgery — * Polyp resection with Hysteroscopic scissors or Versapoint
  * Resection of myoma with Resectoscope Storz or Versapoint
  * Septum resection with Resectoscope Storz or Versapoint
  * Resection of adhesions with Hysteroscopic scissors or Versapoint
  Arms: 2
Drug: Ofloxacinum/Doxycycline — Treatment of endometrial inflammation: Ofloxacinum 400mg/day or Doxycyline 2x100mg on day one, followed by 100mg/day during 8 days.
  Arms: 2

SUMMARY:
This is a comparative, controlled trial to evaluate the impact of treating undetected, asymptomatic, predefined minor uterine cavity abnormalities on the success of IVF treatment.

DETAILED DESCRIPTION:
Introduction- Implantation failure after IVF may be due to endometrial function, embryo quality or a combination of both. The prevalence of minor intracavitary pathology in cases with an apparent normal transvaginal sonography (TVS) observed at hysteroscopy has been recorded to be 25-40%. Treatment of such pathology prior to initiating IVF/ICSI has been advocated without high-quality evidence.

Objective- To evaluate the impact of treating undetected, asymptomatic, predefined minor uterine cavity abnormalities on the success of IVF treatment.

Material & methods- Patients, indicated for their first IVF/ICSI treatment cycle at the UMC Utrecht and AZ-VUB Brussels, initially underwent TVS. In case of a normal TVS these patients were scheduled for hysteroscopy in the early-mid follicular phase of the cycle, one to three months before starting IVF/ICSI treatment. Vaginoscopic hysteroscopy was performed in an ambulatory office setting. During the hysteroscopy a biopsy was taken, to diagnose chronic endometrial inflammation. In case of finding a predefined intra uterine abnormality (polyp, myoma, adhesion, septum, endometrial inflammation) randomisation took place if prior to hysteroscopy informed consent had been obtained for endoscopy treatment versus no treatment. Shortly after the hysteroscopy, IVF/ICSI treatment was initiated and outcome during one year treatment period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Normal Transvaginal Ultrasound
* No prior hysteroscopy
* Regular menstrual cycle
* Single embryo transfer
* BMI between 18 and 29
* Presence of both ovaries
* Primary or secondary infertility
* Women indicated for a first IVF/ICSI cycle

Exclusion Criteria:

* Recurrent miscarriage
* Prior hysteroscopic treatments
* Endometriosis > AFS Stage II
* Meno-metrorrhagia (defined as any intermenstrual loss of blood)
* Submucosal/Intracavitary Fibroids taking more than 50% of the cavity
* Hydrosalpinx
* FSH/LH > 12IU/L on day 3
* Polyps taking more than 50% of the cavity
* Severe adhesions > grade II

Max Age: 36 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 700 (Actual)
Dates: Start 2007-06; Primary Completion 2008-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Cumulative implantation rate | One year

SECONDARY OUTCOMES:
Cumulative ongoing pregnancy | One year
Presence of minor uterine abnormalities | At hysteroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Bart CJM Fauser, Prof. dr., Study Chair — UMC Utrecht; Paul Devroey, Prof. dr., Study Chair — AZ-VUB; Frank JM Broekmans, Dr., Study Director — UMC Utrecht; Human M Fatemi, Dr., Study Director — AZ-VUB; Jenneke C Kasius, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Smit JG, Kasius JC, Eijkemans MJ, Veersema S, Fatemi HM, Santbrink van EJ, Campo R, Broekmans FJ. The international agreement study on the diagnosis of the septate uterus at office hysteroscopy in infertile patients. Fertil Steril. 2013 Jun;99(7):2108-13.e2. doi: 10.1016/j.fertnstert.2013.02.027. Epub 2013 Mar 13. PMID 23499151